CLINICAL TRIAL: NCT01425918
Title: Effects of Self-Generated Experiences on Social Cognitive Development in Young Children With Autism
Brief Title: Social Cognitive Development in Young Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: Autism Speaks (Other)
Responsible Party: Principal Investigator, Rebecca Landa, Principal Investigator, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00050400
Record Dates: First submitted 2011-06-13; First posted 2011-08-30 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; language; social; toddlers
MeSH Terms: conditions — Autism Spectrum Disorder; Language

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Social Enhancement Intervention (Experimental): * For 5 months children will come in 4 days a week for 2-2.5 hours a session to participate in a classroom in an attempt to increase social communication and understanding.
  * Parent education sessions once a week for 2 hours each session over the 5-month period.
  Interventions: Behavioral: Social Enhancement Intervention; Behavioral: Parent Education
- Parent Education (Active Comparator): o Parent education sessions once a week for 2 hours each session over the 5-month period.
  Interventions: Behavioral: Parent Education

INTERVENTIONS:
Behavioral: Social Enhancement Intervention — The intervention will be conducted at our center and focuses on providing an invigorating learning environment in which emerging social skills/knowledge are the focus of intervention with the aim of bringing them to a higher level of maturity, integrated with existing abilities, and used functionally. Learning with and through peers, provides the opportunity to address abnormal peer relationships for developmental level. Providing an enriched environment with toys, structured learning, and opportunities for ongoing engagement we offer the children robust learning experiences. Parent training sessions will focus on strategies aimed at improving child social engagement and communication.
  Arms: Social Enhancement Intervention
Behavioral: Parent Education — Parent education sessions will focus on topics related to autism, learning styles, interventions, and resources. The curriculum provides parents with information about child development and autism as well as instructional strategies (e.g., responsive teaching strategies, principles of applied behavior analysis) for use at home to enhance their children's communication, engagement, and play development. Concrete examples for home-based implementation are presented. Each week, homework will be given and parents will be encouraged to practice the strategies daily at home. No direct coaching to parents during interaction with their children or direct intervention with the child will be provided.

SUMMARY:
Through the development of a novel treatment targeting core Autism Spectrum Disorder (ASD) social deficits and studying the efficacy of this intervention, the investigators hope to provide a means for children with ASD to more effectively and efficiently process social information and enable them to more successfully engage in social interactions. Children between the ages of 24 and 36 months and their families may join.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 24 to 42 months old
* Children must meet criteria for ASD or autism on the ADOS (Lord et al., 2000) plus receive a clinical judgment of PDD-NOS or autism by the study team
* Score ≥ 16 months on the Visual Receptive subtest and ≥ 9 months on the Receptive Language subtest on the Mullen Scales of Early Learning and/or the Vineland Adaptive Behavior Scales at the time of eligibility testing.
* The parent (or other primary caregiver, such as grandparent) in the PE condition must agree to attend the training sessions each week for the 5-month period.
* The parent must agree to bring their child in for testing at all testing points (pre-testing, post-testing, follow-up testing).
* Parents must be between the ages of 18 and 65 years old
* It is not required that English be their primary language, but they must be fluent in English (or if the child is nonverbal he/she must hear English most of the time at home)

Exclusion Criteria:

* <34 weeks or >42 weeks gestational age
* <2500 grams birth weight, severe birth trauma
* Head or serious bodily injury sustained before or during the study
* Illicit drug or excessive alcohol exposure (defined in our telephone screening interview)
* Major hearing or visual impairment
* Non-febrile seizures
* Any known genetic syndrome
* Mitochondrial disorders
* Severe birth defects
* No foster children may participate
* The child must not be adopted
* The child must not be participating in another intervention study simultaneously or be simultaneously enrolled in the CARD clinic's Achievements, Early Achievements, TIPS, Jump Start, or Play with Me programs.
* Unable to provide baseline data on the eye tracking measure at time of pretesting (e.g., tracker unable to read eye movements)
* Has a sibling participating in this study

Ages: 24 Months to 42 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2012-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in Baseline Eye Tracking Tasks | 5 months into treatment and 5 months after the treatment ends
Change in Baseline Communication and Symbolic Behavior Scale Developmental Profile | 5 months into treatment and 5 months after the treatment ends
Change in Baseline Spontaneous Imitation Task | 5 months into treatment and 5 months after the treatment ends

SECONDARY OUTCOMES:
Change in Baseline Autism Diagnostic Observation Schedule | 5 months into treatment and 5 months after the treatment ends
Change in Baseline Mullen Scales of Early Learning | 5 months into treatment and 5 months after the treatment ends
Change in Baseline Action/intention understanding taks | 5 months into treatment and 5 months after the treatment ends

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Landa, PhD, CCC-SLP, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

REFERENCES:
- [Background] Landa RJ, Holman KC, O'Neill AH, Stuart EA. Intervention targeting development of socially synchronous engagement in toddlers with autism spectrum disorder: a randomized controlled trial. J Child Psychol Psychiatry. 2011 Jan;52(1):13-21. doi: 10.1111/j.1469-7610.2010.02288.x. Epub 2010 Dec 3. PMID 21126245
- [Background] Libertus K, Needham A. Teach to reach: the effects of active vs. passive reaching experiences on action and perception. Vision Res. 2010 Dec;50(24):2750-7. doi: 10.1016/j.visres.2010.09.001. Epub 2010 Sep 7. PMID 20828580
- [Background] Sullivan M, Finelli J, Marvin A, Garrett-Mayer E, Bauman M, Landa R. Response to joint attention in toddlers at risk for autism spectrum disorder: a prospective study. J Autism Dev Disord. 2007 Jan;37(1):37-48. doi: 10.1007/s10803-006-0335-3. Epub 2007 Jan 10. PMID 17216332